CLINICAL TRIAL: NCT00193388
Title: Phase II Trial of Weekly Topotecan in the Second-Line Treatment of Small Cell Lung Cancer
Brief Title: Weekly Topotecan in the Second-Line Treatment of Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 66; 104864664
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Topotecan

INTERVENTIONS:
Drug: Topotecan

SUMMARY:
In this phase II trial, we will evaluate the weekly schedule of topotecan in the second-line treatment of patients with small cell lung cancer

DETAILED DESCRIPTION:
Upon determination of eligibility, all patients will be receive:

* Topotecan

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Small Cell Lung cancer
* Progression after one previous regimen
* Measurable or evaluable disease
* Able to perform activities of daily living with assistance
* Adequate bone marrow, liver and kidney function
* No more than three previous courses of radiation therapy
* Accessible for treatment and follow up
* Must give written informed consent prior to study entry

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Central nervous system involvement
* Serious or active infection
* Serious underlying medical condition
* Other active neoplasms

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-09; Primary Completion 2004-12 (Actual); Study Completion 2007-02

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Median survival
1-year survival
Symptomatic improvement

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Greco, MD, Principal Investigator — SCRI Development Innovations, LLC